CLINICAL TRIAL: NCT03705819
Title: Exploratory Evaluation of [11C]-NOP46 Pharmacokinetics With Positron Emission Tomography (PET)
Brief Title: Exploratory Evaluation of [11C]-NOP46
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAQ8138
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain
Keywords: [11C]-NOP46
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Masking Description: Open Label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Experimental): In Stage 1, five healthy volunteers will receive a microdose of [11C]-NOP46 and undergo serial whole body PET/CT scans for up to 240 minutes post-administration. These image sets will be used to evaluate [11C]-NOP46 biodistribution and derive dosimetry estimates.
  Interventions: Drug: [11C]-NOP46; Radiation: PET/CT scan
- Individuals with Focal Pain (Experimental): In Stage 2, up to 30 subjects with focal pain will receive a microdose of [11C]-NOP46 and undergo PET/CT scans for up to 60 minutes in length. The results of Stage 1 will inform the scanning parameters (uptake period, scan length, reconstruction parameters, etc.) for Stage 2.
  Interventions: Drug: [11C]-NOP46; Radiation: PET/CT scan

INTERVENTIONS:
Drug: [11C]-NOP46 — Subjects will receive a microdose (≤10 µg) of [11C]-NOP46.
Radiation: PET/CT scan — After subjects receive a microdose of [11C]-NOP46, whole body PET/CT scan(s) will be performed to determine dosimetry and perform an initial safety evaluation of the radiotracer in Stage 1 and region of interests in Stage 2.

SUMMARY:
This is an open-label, single center design. In the first stage, five (5) healthy individuals will receive a microdose (10µg) of [11C]-NOP46, immediately followed by whole body positron emission tomography (PET)/computed tomography (CT) to determine dosimetry and perform an initial safety evaluation of the radiotracer. If no toxicities develop, then the investigation will move to the second stage, in which thirty (30) patients with chronic pain will receive a microdose of [11C]-NOP46 followed by PET/CT of region of interests.

DETAILED DESCRIPTION:
Pain is a natural response to injury. Pain lets us know there may be damage to our bodies. Pain is the way our body tells us that we must take care of ourselves. Chronic pain is different. Chronic pain is pain that lasts for a long time. Chronic pain can last for weeks, months, and even years. In some cases chronic pain remains without any sign of body damage. Today, there is no way for a doctor to measure someone's chronic pain or accurately determine many details about chronic pain. The investigators at Columbia University are interested in new imaging test that could help doctors look at chronic pain and help patients with chronic pain. The new imaging test uses a new drug called [11C]-NOP46. [11C]-NOP46 is a radioactive drug and is experimental. It is not approved by the Food and Drug Administration (FDA). The investigators believe that, when given to patients, this new drug can go to the exact places of chronic pain within the body. Once the drug goes to the places of chronic pain, a special camera, called a Positron Emission Tomography (PET) camera, can be used to take pictures of the drug. In this study, the investigators will give [11C]-NOP46 to up to 35 subjects.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be 18 years of age or older, able to read, understand, and voluntarily sign an informed consent document.

For Healthy Volunteers:

* Volunteers must have no current medical history of sustained pain from a focal injury.
* Negative pregnancy test if female of childbearing potential.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

Patients with Focal Pain:

* Subjects must have current pain from a focal injury for which they are under a physician's care.
* Subjects must have moderate to severe pain, defined as >4 on the Visual Analogue Scale
* Subjects must have a negative pregnancy test if female of childbearing potential.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Participants with evidence of diffuse pain at the time of enrollment up to agent administration are to be excluded from this study.
* Inability to discontinue pain medication(s) for 48 hours prior to agent administration.(Enrolled participants who have taken pain medication within 48 hours of agent administration may be either withdrawn from the study or rescheduled at the PI's discretion).
* Concomitant medication use (including suspected illicit drugs use) that, in the judgment of the investigator, would make the participant inappropriate for enrollment.
* Severe concurrent disease, infection, or medical co-morbidity that, in the judgment of the investigator, would make the participant inappropriate for enrollment.
* Participants who are receiving any other investigational agents.
* Women who are pregnant or breastfeeding.
* Subjects who are unable to tolerate PET/CT imaging.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Uptake ratio for site with pain is >1 | 48 hours post-scan
  The uptake ratio for the site with pain to the site without pain is greater than 1 in the focal pain subjects

SECONDARY OUTCOMES:
Occurrence of Physiologic Effects of Single Micro-dose of [11C]-NOP46 | 48 hours post-scan
  Total number of physiologic effects associated with a single micro-dose administration of [11C]-NOP46

CONTACTS AND LOCATIONS:
Overall Officials: Akiva Mintz, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Final data analysis and conclusion will be submitted to scientific journals and made available for publication.

REFERENCES:
- [Background] Voscopoulos C, Lema M. When does acute pain become chronic? Br J Anaesth. 2010 Dec;105 Suppl 1:i69-85. doi: 10.1093/bja/aeq323. PMID 21148657
- [Background] Jamison RN, Serraillier J, Michna E. Assessment and treatment of abuse risk in opioid prescribing for chronic pain. Pain Res Treat. 2011;2011:941808. doi: 10.1155/2011/941808. Epub 2011 Oct 11. PMID 22110936
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: overdoses of prescription opioid pain relievers---United States, 1999--2008. MMWR Morb Mortal Wkly Rep. 2011 Nov 4;60(43):1487-92. PMID 22048730
- [Background] Pike VW. PET radiotracers: crossing the blood-brain barrier and surviving metabolism. Trends Pharmacol Sci. 2009 Aug;30(8):431-40. doi: 10.1016/j.tips.2009.05.005. Epub 2009 Jul 16. PMID 19616318
- See also: Centers for Disease Control and Prevention (2011). Prescription painkiller overdoses in the U.S. — https://archive.cdc.gov/#/details?url=https://www.cdc.gov/vitalsigns/painkilleroverdoses/index.html